CLINICAL TRIAL: NCT01533155
Title: A Randomized, 2-Part, Crossover, Single Center Study to Evaluate Effect of Quinidine on the Pharmacokinetics of NKTR-118 and the Concomitant Effect of Quinidine and NKTR-118 on Morphine-induced Miosis
Brief Title: Study in Healthy Volunteers to Investigate the Effects of Quinidine on the Pharmacokinetics of NKTR-118
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D3820C00011
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Drug Induced Constipation
Keywords: Phase 1; Healthy male and female volunteers; Drug-drug interaction; Pharmacokinetics; NKTR-118
MeSH Terms: interventions — Quinidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- NKTR-118/ Quinidine (Active Comparator): One 25-mg NKTR-118 tablet will be administered once with 3 Quinidine 200mg tablets in the morning of period 1 or period 2 (part 1)
  Interventions: Drug: Nektar 118; Drug: Quinidine
- NKTR-118/ Placebo (Placebo Comparator): One 25-mg NKTR-118 tablet will be administered once with 3 Placebo tablets in the morning of period 1 or period 2 (part 1)
  Interventions: Drug: Nektar 118; Drug: Quinidine placebo
- NKTR-118/ Quinidine/ Morphine (Active Comparator): One 25-mg NKTR-118 tablet will be administered with 3 Quinidine 200mg tablets with Morphine inj 5mg/70kg once in the morning on period 3 or period 4 (Part 2)
  Interventions: Drug: Nektar 118; Drug: Quinidine; Drug: Quinidine placebo; Drug: Morphine
- NKTR-118/ Placebo/ Morphine (Placebo Comparator): One 25-mg NKTR-118 tablet will be administered with 3 placebo tables with Morphine inj 5mg/70kg once in the morning of period 3 or period 4 (part 2)
  Interventions: Drug: Nektar 118; Drug: Morphine

INTERVENTIONS:
Drug: Nektar 118 — Oral 25 mg tablet
Drug: Quinidine — Oral 200 mg tablet
  Arms: NKTR-118/ Quinidine; NKTR-118/ Quinidine/ Morphine
Drug: Quinidine placebo — Oral Tablet
  Arms: NKTR-118/ Placebo; NKTR-118/ Quinidine/ Morphine
Drug: Morphine — 10 mg/ml, intravenously
  Arms: NKTR-118/ Placebo/ Morphine; NKTR-118/ Quinidine/ Morphine

SUMMARY:
Study in healthy volunteers to investigate the effects of Quinidine on the Pharmacokinetics of NKTR-118

DETAILED DESCRIPTION:
A Randomized, 2-Part, Crossover, Single Center Study to Evaluate Effect of Quinidine on the Pharmacokinetics of NKTR-118 and the Concomitant Effect of Quinidine and NKTR-118 on Morphine-induced Miosis

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Male and female (nonchildbearing potential, nonlactating) healthy volunteers aged 18 to 55 years inclusive, with suitable veins for cannulation or repeated venipuncture.
* Female volunteers must be nonpregnant and nonlactating. Women of childbearing potential must have negative pregnancy test (screening and admission) and be using a highly-effective form of birth control for 3 months before enrollment.
* Male volunteers should be willing to use barrier contraception ie, condoms, from the first day of dosing until 3 months after dosing with the IP. The female partner should use contraception during this period.
* Volunteers must have a BMI between 18 and 30 kg/m2, inclusive, and weigh at least 50 kg.

Exclusion Criteria:

* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine) which, may put the volunteer at risk of participation in the study, or influence of the ADME of drugs.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IP.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator.
* History (personal or family) of torsades de pointes, any other polymorphic ventricular tachycardia, long QT syndrome, sudden death or Brugada syndrome, or personal history of sustained (greater than 30 s) monomorphic ventricular tachycardia.
* Abnormal vital signs, after 10 minutes supine rest as defined in protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetic (PK) profile for NKTR- 118 in terms of maximum observed plasma concentration (Cmax), time to Cmax (tmax), apparent terminal half-life (t1/2λz). | At predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose.
Description of the PK profile for NKTR- 118 in terms of apparent terminal rate constant (λz), area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC). | At predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose.
Description of the PK profile for NKTR 118 in terms of area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-t)]. | At predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose.
Description of the PK profile for NKTR 118 in terms of area under the plasma concentration-time curve from time zero to 24 hours [AUC(0-24)]. | At predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose.
Description of the PK profile for NKTR 118 in terms of apparent oral clearance from plasma (CL/F), and apparent volume of distribution during the terminal phase (Vz/F). | At predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose.

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events, clinical laboratory assessments , vital signs (blood pressure and pulse rate), physical examinations, electrocardiograms and Columbia-Suicide Severity Rating Scale. | From baseline up to 21 days.
Description of results from pupillary measurements in terms of size change from baseline on both eyes in mm. (Measurements in 4 different conditions: dark, 0.04 lux, 0.4 lux and 4 lux) | Measurments from baseline day -1, and at 0.5, 1, 2, 3, 4, 6, and 24 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Leese, MD, Principal Investigator — Quintiles Kansas United states; Mark Sostek, MD, Study Director — Astrazeneca, Wilmington US; Bo Fransson, MD, Study Chair — Astrazeneca, Sodertalje Sweden
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: Clinical_Study_Report_Synopsis_D3820C00011 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1393&filename=Clinical_Study_Report_Synopsis_D3820C00011.pdf